CLINICAL TRIAL: NCT02019992
Title: Plasma Levels of Mitochondrial DNA in Patients Presenting to ICU With Sepsis
Brief Title: Investigation of Plasma Mitochondrial DNA Level in Septic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, lemeng zhang, md, Central South University
Other Study IDs: CSU-ICU-2013-01
Record Dates: First submitted 2013-12-12; First posted 2013-12-24 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Sepsis; Inflammation
Keywords: sepsis; mitochondrial DNA; systemic inflammation; outcome
MeSH Terms: conditions — Sepsis; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- sepsis: sepsis defined as suspected infection and systemic inflammatory response
- severe sepsis: sepsis with organ dysfunction or septic shock defined as sepsis plus hypotension
- control group: control defined as non-infected patients without systemic inflammatory response.

SUMMARY:
To determine the plasma levels of mtDNA in ICU department patients with and without sepsis and evaluate their association with severity, systemic inflammation and outcomes. Plasma from control, septic and severe septic patients will be collected. The level of mtDNA and systemic cytokine will be measured.

DETAILED DESCRIPTION:
Clinical protocol:

Patients were enrolled into one of three cohorts: (i) sepsis defined as suspected infection and systemic inflammatory response, (ii) septic shock defined as sepsis plus hypotension, and (iii) control defined as non-infected patients without systemic inflammatory response.

Methods:

Plasma levels of mtDNAs were measured using real-time quantitative polymerase chain reaction. Levels of mtDNAs were compared among each group, and linear regression was used to assess the association between mtDNAs, IL-6, TNF a and IL-1b in patients with sepsis. The correlation between plasma mtDNA and severity, systemic inflammation and outcomes will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sepsis and severe sepsis was according to the following guild-line. "Surviving Sepsis Campaign: International Guidelines for Management of Severe Sepsis and Septic Shock: 2012"

Exclusion Criteria:

* Patients lost following-up. Patients who refuse to sign the consent form.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sepsis and severe septic patients enrolled in 2014 will be collected.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-01 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
change from baseline in plasma mtDNA in septic patients at 7 days | 7 days
  The change from baseline in plasma mtDNA in septic patients at 7 days will be measured by real-time PCR.

SECONDARY OUTCOMES:
change from baseline in plasma IL-6, TNF a and IL-1b level in septic patients at 7 days | 7 days
  The change from baseline in plasma IL-6, TNF a and IL-1b level in septic patients at 7 days will be measured by ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: lemeng zhang, md, Principal Investigator — Central South University
Locations (1):
- Xiangya Hospital, Changsha, Hunan, China